CLINICAL TRIAL: NCT06137508
Title: Cancer-associated Cachexia in Patients With Incurable Gastroesophageal Cancer
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Rikke Krabek, MD, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-23050300
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Gastro-Esophageal Cancer
Keywords: Cancer; Cancer Cachexia; Sarcopenia; Neoplasms; Metabolism
MeSH Terms: conditions — Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with incurable gastroesophageal cancer are at high risk of cancer cachexia with an estimated prevalence of 60-80%. Cancer cachexia is defined as ongoing loss of skeletal muscle mass with or without loss of fat mass and is associated with impaired quality of life, loss of physical function, treatment intolerability, and increased mortality.

Cancer cachexia is a multifactorial syndrome, and in patients with gastroesophageal cancer, the wasting is compounded by a high prevalence of dysphagia. To date, no drug therapy has been approved for the treatment for cancer cachexia. Sufficient nutritional support is imperative in cachexia treatment, but to effectively treat cancer cachexia there is a need to fully understand the biological mechanisms underpinning the wasting syndrome.

The primary objective of the present cohort study is to determine the incidence and extend of skeletal muscle wasting in patients with incurable gastroesophageal cancer. The investigators will also investigate the prevalence of low skeletal muscle at time of diagnosis. The secondary objective is to investigate, if loss of skeletal muscle is associated with treatment intolerance and increased mortality.

Furthermore, the investigators aim to explore factors differentially expressed in the circulation, in skeletal muscle, and in adipose tissue of patients experiencing wasting compared with patients not experiencing wasting.

The study is a prospective cohort study including patients with incurable gastroesophageal cancer referred to first line chemotherapy. Blood and plasma samples as well as clinical and simple functional assessments will be obtained from all patients. The participants will also be offered to take part in a sub-study in which, we will collect skeletal muscle and subcutaneous adipose tissue.

The main questions the investigators aim to answer are:

* What is the prevalence and extent of skeletal muscle mass wasting in patients with incurable gastroesophageal cancer?
* Are the loss of skeletal muscle mass and low skeletal muscle mass associated with treatment intolerability and overall survival in patients with incurable gastroesophageal cancer?
* Can there be identified potential biological processes and factors in skeletal muscle, adipose tissue, and plasma that contribute to the loss of skeletal muscle mass in patients with incurable gastroesophageal cancer?

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for participation are any patient diagnosed with histologically verified, incurable cancer of the esophagus, stomach, or gastroesophageal junction, referred to first line chemotherapy.

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with histologically verified, incurable cancer of the esophagus, stomach, or gastroesophageal junction, referred to first line chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle area | Baseline, 9 and 18 weeks
  CT assessed changes in skeletal muscle index at L3 (cm2/m2)

SECONDARY OUTCOMES:
Cancer-specific survival | Until 3 years after inclusion
  Proportion of patients who have not died from gastroesophageal cancer.
Over-all survival | 1, 2, and 3 years after inclusion
  Proportion of patients who have not died.
Progression-free survival | 1, 2, and 3 years after inclusion
  Time to progression.
Treatment tolerance: Hospitalization | Baseline, 9 and 18 weeks
  Unscheduled hospitalization
Treatment tolerance: Relative dose intensity | Baseline, 9 and 18 weeks
  Treatment tolerance assessed by the delivery of chemotherapy (relative dose intensity)
Treatment tolerance: Number of series received | Baseline, 9 and 18 weeks
  Treatment tolerance assessed by the delivery of chemotherapy (number of series received)
Treatment tolerance: Tolerated dose | Baseline, 9 and 18 weeks
  Treatment tolerance assessed by the delivery of chemotherapy (dose reduction)
Treatment tolerance: Permanent discontinuation of the treatment | Baseline, 9 and 18 weeks
  Treatment tolerance assessed by the delivery of chemotherapy (permanent discontinuation of the treatment)
Muscle strength: Hand grip strength | Baseline, 9 and 18 weeks
  Changes in hand grip strength, assessed using a dynamometer
Functional performance: Sit-to-stand | Baseline, 9 and 18 weeks
  Changes in sit-to-stand power

OTHER OUTCOMES:
Molecular factors associated with changes in skeletal muscle mass | Baseline, 9 and 18 weeks
  Explorative analysis of molecular factors expressed in plasma, skeletal muscle- and adipose tissue associated with changes in skeletal muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Casper Simonsen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No